CLINICAL TRIAL: NCT07378371
Title: Proactive Temperature Management and Delirium After Cytoreductive Surgery With HIPEC: A Randomized Controlled Trial
Brief Title: Proactive Temperature Management in CRS-HIPEC for Prevention of Delirium
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aerospace Center Hospital (Other)
Responsible Party: Principal Investigator, Xinrui Yin, Principal Investigator, Aerospace Center Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XYin-HIPEC-2026-01
Record Dates: First submitted 2026-01-18; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pseudomyxoma Peritonei; Postoperative Delirium (POD)
Keywords: Cytoreductive Surgery; HIPEC; Hyperthermic Intraperitoneal Chemotherapy; Temperature Management; Goal-Directed Therapy
MeSH Terms: conditions — Pseudomyxoma Peritonei; Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDTM Group (Experimental): Participants assigned to this group receive a protocolized, phase-based temperature management algorithm. This includes strict normothermia maintenance during cytoreduction, anticipatory pre-cooling prior to HIPEC perfusion, and proactive cooling during the hyperthermic phase to attenuate thermal variability .
  Interventions: Procedure: Proactive Goal-Directed Temperature Management
- Usual Care Group (Active Comparator): Participants receive standard institutional thermal management characterized by a reactive approach. Therapeutic interventions (warming or cooling) are determined by the attending anesthesiologist based on observed threshold violations (e.g., core temperature <36.0°C or >38.5°C) rather than a prespecified goal-directed algorithm .
  Interventions: Procedure: Standard Reactive Temperature Management

INTERVENTIONS:
Procedure: Proactive Goal-Directed Temperature Management — The protocol consists of four phases:
  Cytoreductive Phase: Maintain core temperature 36.5-37.5°C.
  Pre-cooling Phase: Initiated ~30 min before HIPEC (e.g., during closure), targeting 36.0-36.3°C.
  HIPEC Phase: Proactive cooling to target 37.5-38.0°C; escalation triggered at 37.8°C. 4. Rewarming Phase: Restore 36.5-37.5°C prior to ICU transfer .
  Arms: GDTM Group
Procedure: Standard Reactive Temperature Management — Hypothermia Management: Active warming initiated reactively only when core temperature falls below 36.0°C.
  Pre-cooling: No anticipatory pre-cooling is performed. 3. HIPEC Phase: Active cooling withheld unless core temperature exceeds standard safety thresholds (typically >38.5°C) or for immediate safety indications .
  Arms: Usual Care Group

SUMMARY:
This randomized controlled trial evaluates the efficacy of a proactive Goal-Directed Temperature Management (GDTM) protocol in reducing postoperative delirium among patients undergoing Cytoreductive Surgery (CRS) with Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for pseudomyxoma peritonei.

CRS-HIPEC presents a unique physiological challenge characterized by a biphasic thermal trajectory: potential hypothermia during extensive surgery followed by rapid iatrogenic hyperthermia during perfusion. This study compares a standardized GDTM strategy-which incorporates strict normothermia maintenance and anticipatory pre-cooling prior to perfusion-against standard reactive thermal management. The primary objective is to determine if optimized thermoregulation can attenuate thermal variability and improve early neurocognitive recovery.

DETAILED DESCRIPTION:
Cytoreductive surgery (CRS) combined with hyperthermic intraperitoneal chemotherapy (HIPEC) imposes a formidable physiologic burden, involving extensive resections and a distinctive thermal paradox. Patients typically experience a prolonged cytoreductive phase prone to inadvertent hypothermia, followed by protocol-driven hyperthermia during the perfusion phase. This rapid thermal fluctuation may disrupt blood-brain barrier integrity and amplify neuroinflammation, potentially contributing to postoperative delirium (POD).

Despite these risks, perioperative thermoregulation often remains reactive, with interventions initiated only after temperature thresholds are violated. Evidence-based recommendations for managing the iatrogenic heat load inherent to HIPEC remain undefined.

This single-center, parallel-group, randomized controlled trial aims to address this gap. Eligible adult patients scheduled for elective CRS-HIPEC are randomized to receive either proactive Goal-Directed Temperature Management (GDTM) or Usual Care. The GDTM protocol utilizes a phase-based algorithm, including specific targets for normothermia during resection and a "thermal buffer" created by anticipatory cooling prior to the hyperthermic phase. The Usual Care group receives standard reactive management where interventions are triggered primarily by observed threshold violations.

The primary endpoint is the incidence of POD within the first 7 postoperative days. Secondary endpoints include delirium-free days, intraoperative thermal exposure metrics, delayed neurocognitive recovery, and 30-day major complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18-80 years).

American Society of Anesthesiologists (ASA) physical status of I to III.

Scheduled for elective Cytoreductive Surgery (CRS) with Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for Pseudomyxoma Peritonei (PMP).

Written informed consent obtained from the participant or legally authorized representative.

Exclusion Criteria:

* Known diagnosis of dementia, major neurocognitive disorder, or severe psychiatric illness (e.g., schizophrenia) documented in the medical record.

Acute central nervous system pathology likely to confound delirium assessment (e.g., recent stroke, active seizure disorder, or traumatic brain injury).

Severe sensory or language barriers precluding valid cognitive screening (e.g., profound deafness or blindness, or language barriers not correctable with translation).

Preoperative coma, mechanical ventilation, or deep sedation precluding reliable baseline assessment.

Emergency surgery or repeat CRS-HIPEC during the same hospital admission.

History of alcohol or substance abuse likely to precipitate withdrawal symptoms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Delirium | From ICU admission through postoperative day 7 (or hospital discharge, whichever occurs first)
  Delirium is assessed twice daily (08:00-10:00 and 18:00-20:00) using the Confusion Assessment Method for the ICU (CAM-ICU) for mechanically ventilated or ICU patients, and the standard CAM for ward patients. Postoperative delirium is defined as at least one positive CAM-ICU or CAM assessment during the assessment window .

SECONDARY OUTCOMES:
Delirium- and Coma-Free Days (DCFDs) | Within 7 days postoperatively
  Calculated as the number of days alive and free of both delirium and coma. A day is scored as "free" only if the patient is alive, not comatose, and delirium-negative on all assessments .
Intraoperative Thermal Exposure (AUC >38.5°C) | From the initiation of HIPEC perfusion until the completion of perfusion, approximately 90 minutes.
  Calculated as the Area Under the Curve (AUC) for core temperature >38.5°C during the HIPEC phase to quantify physiologic thermal load.
30-Day Major Complications Composite | Within 30 days postoperatively
  A composite of Clavien-Dindo grade III-V complications (including mortality).
Delayed Neurocognitive Recovery (DNR) | Discharge (or postoperative day 7) and 1 month postoperatively
  Assessed using the Montreal Cognitive Assessment (MoCA). DNR is defined as a decline in MoCA score of ≥1 SD from the preoperative baseline mean, adjusted for age and education .
Quality of Recovery (QoR-15 Score) | Postoperative days 1, 3, and 7
  Evaluated using the QoR-15 questionnaire, a 15-item patient-reported outcome measure. Scores range from 0 to 150, with higher scores indicating better quality of recovery.
Postoperative Pain Intensity (NRS Score) | Postoperative days 1, 2, and 3
  Assessed using an 11-point Numeric Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst pain imaginable.
Length of Stay (ICU and Hospital) | From date of surgery until date of hospital discharge, assessed up to 30 days.
  Duration of stay in the Intensive Care Unit (ICU) and total hospital length of stay from surgery to discharge
Cumulative Opioid Consumption | From the end of surgery up to 72 hours postoperatively.
  Total postoperative opioid consumption converted to morphine milligram equivalents (MME).
Incidence of Severe Thermal Excursions | From the start of anesthesia induction until the end of surgery, approximately 10 hours
  Defined as core temperature <35.0°C (severe hypothermia) or >39.0°C (severe hyperthermia)
Incidence of Thermal-Related Adverse Events | From the end of surgery until hospital discharge, assessed up to 30 days.
  Includes postoperative shivering requiring pharmacologic treatment and device-related skin injury (e.g., thermal burns, cold injury, pressure ulcers).

CONTACTS AND LOCATIONS:
Overall Officials: Xiangli Zheng, Study Chair — Aerospace Center Hospital
Locations (1):
- Aerospace Center Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided